CLINICAL TRIAL: NCT06589245
Title: The Safety and Toxicity of Inhaled Ciclesonide (i.e., Alvesco) in Preterm Infants at Risk for Developing Bronchopulmonary Dysplasia
Brief Title: Inhaled Ciclesonide Study in Preterm Infants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Venkatesh Sampath (Other)
Collaborators: University of Pittsburgh (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor-Investigator, Venkatesh Sampath, Physician-Scientist, Children's Mercy Hospital Kansas City
Organization: Children's Mercy Hospital Kansas City (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00003195; R21HD116421 (NIH)
Record Dates: First submitted 2024-08-20; First posted 2024-09-19 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Bronchopulmonary Dysplasia
MeSH Terms: conditions — Bronchopulmonary Dysplasia | interventions — ciclesonide

STUDY DESIGN:
Intervention Model Description: An open label dose escalation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ciclesonide (Experimental): Eligible infants will be approached by study team. Parents whose infants consent to the study drug will enter the dose-escalation part of the study. Inhaled Alvesco will be administered daily for 14 days at escalating doses 80mcg and 160mcg.
  Interventions: Drug: Alvesco Inhalant Product
- Control (No Intervention): Eligible infants will be approached by study team. Parents who refuse consent to the study drug will have standard of care. These parents can accept for their infant's de-identified clinical data to be used as part of the control group.

INTERVENTIONS:
Drug: Alvesco Inhalant Product — Inhaled Alvesco will be administered daily for 14 days at escalating doses of 80mcg and 160mcg.
  Other Names: ciclesonide
  Arms: Ciclesonide

SUMMARY:
Our overall objective is to conduct a safety study with inhaled ciclesonide to evaluate known glucocorticoids (sGC)-related acute and intermediate toxic effects while measuring for the first time in neonates its systemic absorption and potential bioactivity (i.e. activation of primary target, the GR, in blood cells).

DETAILED DESCRIPTION:
Preterm infants born before 30 weeks gestation are at increased risk of developing bronchopulmonary dysplasia (BPD), a leading cause of death and long-term pulmonary insufficiency. Both hydrocortisone and synthetic glucocorticoids (sGC) are commonly used to prevent BPD in premature infants. Clinical trials have shown that hydrocortisone targeted to infants with emerging lung disease does not prevent BPD, while inhaled sGC therapy has shown mixed efficacy in clinical trials. Dexamethasone (DEX) has been shown in clinical trials to reduce BPD rates in premature infants but is associated with short term and long-term adverse effects including cerebral palsy. There is an unmet need for efficacious Glucocorticoid (GC) therapy in premature infants to prevent BPD without encumbering serious adverse events. To address this challenge, our group has been investigating ciclesonide (CIC), a sGC pro-drug that in the inhaled form is FDA approved for use in asthma and allergic rhinitis in older children. Our published and ongoing work has shown that DEX and CIC regulate GR transcriptional targets and several genes implicated in lung protective effects in neonatal rats. Remarkably, CIC does not suppress somatic growth nor IGF-1 levels, induce hyperglycemia, or cause neuroanatomical changes in the cerebral cortex of neonatal rats, which are known pathologies caused by DEX in premature infants. Furthermore, ongoing studies reveal that CIC is as efficacious as DEX in preventing lung injury in a hyperoxia-model of experimental BPD. This study tests the hypothesis that CIC will have minimal systemic absorption and a favorable safety profile in premature infants at risk of developing BPD.

The fear of long-term neurological adverse effects has limited optimal use of sGC therapy to prevent BPD. This application is significant as it proposes to repurpose CIC, an existing sGC, for novel therapeutic use in preterm infants to prevent BPD. CIC is already FDA-approved for use in children >5 years for allergic rhinitis and asthma, and can be used on a compassionate basis down to 2 years of age. The investigators believe our study is impactful and translationally relevant as it addresses an unmet need for efficacious GC therapy to prevent BPD in premature infants without encumbering the neurological and somatic adverse effects. Successful testing of our hypothesis will pave the way for a large, multicenter randomized control trial of CIC therapy in premature infants to prevent BPD.

ELIGIBILITY:
Inclusion Criteria:

* Viable Infants born between 23 0/7 - 29 6/7 gestation
* Requiring invasive (through an endotracheal tube) mechanical ventilation
* Between day of life 8 to 28.
* Infants have not received dexamethasone for 120 hours
* If receiving hydrocortisone, then receiving ≤ 1mg/kg/day

Exclusion Criteria:

* Infants with major congenital lung or other organ anomalies, life-threatening illness, active sepsis or NEC, and grade IV hemorrhage will be excluded.
* Infants receiving DEX therapy will be excluded.
* We will exclude infants who have had ≥ 1 glucose level > 150mg in the 24 hours prior to study entry or those on insulin therapy to treat hyperglycemia. We will exclude infants who have hypertension (>95% centile for gestational age) in the 48 hours prior to study entry.
* For small for gestational age, we will exclude infants with a birthweight < 5% centile for gestational age.
* Infants with history of recent pulmonary hemorrhage (within 72 hours of study entry) will also be excluded.
* Infants receiving or have received any dexamethasone in the prior 120 hours.
* Infants receiving >1mg/kg/day of hydrocortisone.
* Infants receiving any other inhaled or systemic steroid.

Ages: 8 Days to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2025-09-16 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Number of hyperglycemia events (blood glucose >150mg/dL) during treatment. | Through study completion, an average of 4 months.
  Blood Glucose (BG) levels will be collected 24 hours prior to initiation of study drug and then every 12 hours after initiation of study drug for 2 weeks. BG will be monitored daily for a week after cessation of drug treatment and as per NICU protocol thereafter.
Average change in z-scores for weight, length, and head circumference. | Through the time of discharge, an average of 4 months.
  Baseline weight, head circumference, and length measurements will be measured as per routine NICU standards, which is daily weights and weekly length and head circumference. Weights, lengths and weights/lengths are routinely plotted in the growth chart for each baby in the NICU, and z-scores trajectories deviations (positive or negative) derived against published reference standards for this population. We will compare the average z-score deviations for growth parameters among infants exposed to the study drug and controls unexposed to study drug.
Number of high systolic blood pressure events defined as >95% centile for gestational age and day of life. | Through the time of discharge, an average of 4 months.
  Blood Pressure will be collected 48 hours prior to initiation of study drug as per NICU protocol (at least twice a day) and then every 8 hours after initiation of study drug for 2 weeks. Blood pressure will also be monitored at least daily for first two weeks after cessation of drug treatment, and as per NICU protocol till discharge (at least once a day). Blood pressure is usually monitored using appropriate BP cuff size for weights. If indwelling arterial catheters are present, then blood pressures will be measured that way.
Number of infants who do not pass the Adrenocorticotrophic Hormone (ACTH) stimulation test. | 6 weeks or later after last postnatal steroid course, prior to discharge
  Measured via Adrenocorticotropic Hormone (ACTH) Stimulation Test, which quantifies the increase in cortisol after ACTH administration.
Number of episodes of bronchospasm related to inhaled ciclesonide administration. | The entire duration of the study drug treatment (14 days).
  The investigators will quantify any episodes of bronchospasm as evaluated by changes in oxygenation/ventilation status, auscultation for wheezes and changes in ventilator loops. This is evaluated by experienced respiratory therapists and bedside nurses.
Number of infants who develop oral thrush that require treatment. | The duration of study drug treatment (14 days).
  Bedside nurses routinely evaluate for this common, mostly benign complication of prematurity. We will collect data on % of infants who develop oral thrush and % of infants that require topical treatment among infants exposed to inhaled ciclesonide and the control group.
Compare rates of BPD and severe BPD between cases and controls. | BPD and severe BPD are ascertained at 36 weeks post-menstrual age.
  Investigators will collect and report data on BPD and severity on each infant in the study irrespective of whether they were treated with inhaled ciclesonide or served as a control. We will also compare rates of BPD and severe BPD among the two groups.
Systemic Absorption of inhaled Ciclesonide | Day 1, 3, 7, 15 of study (during drug administration).
  Investigators will measure serum levels of ciclesonide and its active metabolite, des-ciclesonide 3 hour after inhaled drug administration (based on T1/2 in prior studies in children) in peripheral blood by mass spectrometry. This will provide us information on CIC to des-CIC conversion in preterm neonates, as well correlation with doses administered. Measured in picomol/ml (pmol/mL).

SECONDARY OUTCOMES:
Compare rates of extubation success between infants exposed to study drug and controls receiving standard NICU clinical care | Extubation rates will be calculated from the day of study drug initiation to 7 days after cessation of study drug, i.e., a 21 day window.
  Investigators will compare the rates of extubation (weaning from invasive endotracheal tube-delivered mechanical ventilation to nasal respiratory support) between infants receiving study drug and controls not receiving study drug. Successful extubation will be considered as staying extubated for 72 hours.
Assess changes in lung injury and need in mechanical ventilation support. | Baseline, and daily from study drug initiation to 1 week after study drug cessation.
  Lung injury is difficult to characterize in preterm neonates. The pulmonary severity score that combines level and type of support (high frequency oscillator vs. conventional ventilator), oxygen requirements and respiratory drug therapy to calculate a score is accepted as a measure of lung injury and lung disease severity in this population. We will measure pulmonary severity scores to assess lung injury and lung disease severity. Temporal trends will assess whether PSS decreased after initiation of CIC therapy. Higher score indicate a worse outcome. PSS scores range between 0.21 to 2.95

CONTACTS AND LOCATIONS:
Overall Officials: Venkatesh Sampath, MD, Principal Investigator — Children's Mercy Hospital Kansas City; Venkatesh Sampath, MD, Principal Investigator — Physician-Scientist
Locations (1):
- Children's Mercy Kansas City, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No